CLINICAL TRIAL: NCT01201343
Title: Evaluation of Emotional Disorders During Treatment by Interferon Beta in Relapsing-remitting Multiple Sclerosis Patients
Acronym: SEPTIME
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Serono S.A.S, France (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMP 25206
Record Dates: First submitted 2010-09-13; First posted 2010-09-14 (Estimated); Results first posted 2012-04-11 (Estimated); Last update posted 2013-12-27 (Estimated); Status verified 2013-12

CONDITIONS: Multiple Sclerosis, Relapsing, Remitting
Keywords: Multiple sclerosis, relapsing, remitting; Interferon-beta
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Interferon beta-1a

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Interferon beta-1a
  Other Names: Rebif

SUMMARY:
This study is planned to evaluate emotional disorders during treatment by interferon (IFN) beta in relapsing remitting multiple sclerosis (RRMS) subjects. This is an open-label exploratory study with no change of therapeutic behavior but with standardized neuropsychologic follow-up.

DETAILED DESCRIPTION:
This study is planned to evaluate emotional disorders during treatment by IFN beta in RRMS subjects. This is an open-label, prospective, interventional, multicentric study with no change of therapeutic behavior but with standardized neuropsychologic follow-up. Subjects will undergo 13 evaluations (categorical and dimensional evaluations), 3 evaluations will be performed before the treatment (Baseline, Day 7 and 15) and 10 evaluations after the treatment (Month 1, 2, 3, 4, 5, 6, 9, 12, 18 and 24).

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged ≥ 18 years
* Subjects with RRMS
* Subjects with at least 2 relapses in the past two years (with last relapse finished or finishing)
* Subjects with indication of IFN beta treatment determined by the investigator
* Other protocol-defined inclusion criteria may apply

Exclusion Criteria:

* Subjects with secondary progressive multiple sclerosis (MS) without relapse
* Subjects with ongoing acute relapse
* Subjects already being treated with interferon
* Subjects with corticoid therapy for less than 15 days
* Subjects presenting acute major depression or treated with anti-depressant therapy
* Subjects involved in another therapeutic study
* Subjects with any condition which could interfere with a good compliance of this study
* Other protocol-defined exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2005-01; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Brochet, MD, Prof., Principal Investigator — Hôpital PELLEGRIN, Place Amélie Raba Léon 33076 BORDEAUX Cedex

REFERENCES:
- [Background] Radat F, Lafittau M, Ouallet JC, Brochet B, Jouvent R. [Validation of EHD self questionnaire in multiple sclerosis]. Encephale. 2007 Jan-Feb;33(1):49-57. doi: 10.1016/s0013-7006(07)91558-4. French. PMID 17457294
- [Background] Sharrack B, Hughes RA. The Guy's Neurological Disability Scale (GNDS): a new disability measure for multiple sclerosis. Mult Scler. 1999 Aug;5(4):223-33. doi: 10.1177/135245859900500406. PMID 10467380
- [Background] Spielberger, C. D., Gorsuch, R. L., Lushene, R., Vagg, P. R., & Jacobs, G. A. (1983). Manual for the State-Trait Anxiety Inventory. Palo Alto, CA: Consulting Psychologists Press
- [Background] Radloff LS. The CES-D scale: A self-report depression scale for research in the general population. Applied Psychological Measurement. 1977;1:385-401.
- [Background] Spielberger CD. Manual for the State-Anger Expression Inventory. Odessa, FL: Psychological Assessment Resources; 1996

RESULTS

PARTICIPANT FLOW:
Groups:
- Interferon-beta: Participants received interferon-beta based on investigator's discretion as per the clinical practice for 2 years.
Period: Overall Study
Arm/Group | Interferon-beta
Started | 79
Treated | 76
Completed | 60
Not Completed | 19
Not completed — Adverse Event | 6
Not completed — Withdrawal by Subject | 5
Not completed — Lost to Follow-up | 2
Not completed — Lack of Efficacy | 2
Not completed — Participant wrongly included in trial | 1
Not completed — Randomized, not treated | 3

BASELINE CHARACTERISTICS:
Arm/Group | Interferon-beta
Number analyzed (Participants) | 70
Age, Continuous [Mean (Standard Deviation); unit: years] — Out of a total of 79 participants, data for baseline measure (age) was available for 70 participants with at least one interferon-beta intake and with at least one evaluation of the primary criterion.
  years | 37.0 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Out of a total of 79 participants, data for baseline measure (gender) was available for 70 participants with at least one interferon-beta intake and with at least one evaluation of the primary criterion.
  Participants
    Female | 56
    Male | 14

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Emotional Dyscontrol Sub-score of the Depressive Mood Scale (Echelle d'Humeur Depressive [EHD]) Scale at Month 12
Description: EHD scale is a tool to assess the depressive mood dimensions 'lack of emotional control' (emotional dyscontrol) and 'blunted effect' which comprises of 11 items graded in 4 degrees from 1 (not at all) to 4 (very much), where 4 corresponds to the worst state. The emotional dyscontrol sub-score is the sum of items 1, 2, 4, 5, 9, 10, and 11. The total possible score range from 1 (not at all) to 28 (very much), where 28 corresponds to worst state. (Radat F et al., 2007)
Time Frame: Baseline and Month 12
Population: Intent-to-treat (ITT) population: all participants with at least 1 interferon-beta intake and 1 evaluation of primary criterion, that is, at least 1 evaluation before treatment initiation and after Day 0 for emotional dyscontrol sub-score. 'n' signifies those participants who were evaluated for this measure at that time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Interferon-beta
Number analyzed (Participants) | 70
units on a scale
  Baseline (n= 70) | 12.7 (4.4)
  Change at Month 12 (n= 57) | -0.5 (4.2)

2. Primary Outcome: Change From Baseline in Emotional Dyscontrol Sub-score of the EHD Scale at Month 18
Description: as for outcome 1
Time Frame: Baseline and Month 18
Population: ITT population: all participants with at least 1 interferon-beta intake and 1 evaluation of primary criterion, that is, at least 1 evaluation before treatment initiation and after Day 0 for emotional dyscontrol sub-score. 'N' (number of participants analyzed) signifies those participants who were evaluated for this measure at that time-point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Interferon-beta
Number analyzed (Participants) | 61
units on a scale | -0.6 (4.6)

3. Primary Outcome: Change From Baseline in Emotional Dyscontrol Sub-score of the EHD Scale at Month 24
Description: as for outcome 1
Time Frame: Baseline and Month 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Interferon-beta
Number analyzed (Participants) | 63
units on a scale | -0.1 (5.2)

4. Secondary Outcome: Change From Baseline in Emotional Abrasion Sub-score of the EHD Scale at Months 1, 2, 3, 4, 5, 6, 9, 12, 18 and 24
Description: EHD scale is a tool to assess the depressive mood dimensions 'lack of emotional control' (emotional dyscontrol) and 'blunted effect' which comprises of 11 items graded in 4 degrees from 1 (not at all) to 4 (very much), where 4 corresponds to the worst state. The emotional abrasion sub-score is the sum of items 3, 6, 7, and 8. The total possible score range from 1 (not at all) to 16 (very much), where 16 corresponds to worst state. (Radat F et al., 2007)
Time Frame: Baseline, Months 1, 2, 3, 4, 5, 6, 9, 12, 18 and 24
Population: ITT population: all participants with at least 1 interferon-beta intake and 1 evaluation of primary criterion, that is, at least 1 evaluation before treatment initiation and after Day 0 for emotional dyscontrol sub-score. 'n' signifies those participants who were evaluated for this measure at that time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Interferon-beta
Number analyzed (Participants) | 70
units on a scale
  Baseline (n= 70) | 5.6 (1.6)
  Change at Month 1 (n= 64) | 0.3 (1.6)
  Change at Month 2 (n= 62) | -0.1 (1.7)
  Change at Month 3 (n= 64) | -0.0 (1.6)
  Change at Month 4 (n= 59) | -0.0 (1.8)
  Change at Month 5 (n= 58) | -0.2 (1.5)
  Change at Month 6 (n= 56) | -0.3 (1.8)
  Change at Month 9 (n= 58) | -0.1 (1.8)
  Change at Month 12 (n= 57) | -0.0 (2.3)
  Change at Month 18 (n= 61) | -0.3 (1.9)
  Change at Month 24 (n= 63) | -0.3 (1.7)

5. Secondary Outcome: Change From Baseline in State-trait Anxiety Inventory (STAI State) Score at Months 1, 2, 3, 4, 5, 6, 9, 12, 18 and 24
Description: STAI state scale is an auto-evaluation scale for anxiety. This scale includes 20 items that allow quantifying feeling of apprehension, tension, nervousness and worry that the participant feels at the time of the completion of the questionnaire. The 20 items are graded from 1 (no) to 4 (yes), where 'yes' corresponds to the best state for items 1, 2, 5, 8, 10, 11, 15, 16, 19, 20 (scoring was reversed before calculation of total score); and to the worst state for items 3, 4, 6, 7, 9, 12, 13, 14, 17, 18. The total score ranged from 1 (best state) to 80 (worst state). (Spielberger CD et al., 1983)
Time Frame: Baseline, Months 1, 2, 3, 4, 5, 6, 9, 12, 18 and 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Interferon-beta
Number analyzed (Participants) | 70
units on a scale
  Baseline (n= 70) | 35.9 (11.8)
  Change at Month 1 (n= 65) | 0.8 (10.5)
  Change at Month 2 (n= 62) | 0.3 (12.3)
  Change at Month 3 (n= 64) | -1.7 (11.5)
  Change at Month 4 (n= 59) | -1.5 (11.0)
  Change at Month 5 (n= 58) | -0.8 (9.2)
  Change at Month 6 (n= 55) | -1.4 (11.5)
  Change at Month 9 (n= 58) | -0.2 (10.5)
  Change at Month 12 (n= 57) | -0.3 (12.7)
  Change at Month 18 (n= 61) | -1.2 (11.2)
  Change at Month 24 (n= 63) | -1.4 (13.1)

6. Secondary Outcome: Change From Baseline in Center for Epidemiologic Studies Depression (CES-D) Score at Months 1, 2, 3, 4, 5, 6, 9, 12, 18 and 24
Description: CES-D is an auto-questionnaire including 20 items to screen for depressive feelings and behaviour. The 20 items of this scale are graded from 0 (never) to 3 (always), where 3 corresponds to the most severe state with the exception of items 4, 8, 12 and 16 (scoring was reversed before the calculation of the total score). Total score ranged from 0 (never) to 60 (always), where 60 corresponds to most severe state. (Radloff LS, 1977)
Time Frame: Baseline, Months 1, 2, 3, 4, 5, 6, 9, 12, 18 and 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Interferon-beta
Number analyzed (Participants) | 70
units on a scale
  Baseline (n= 70) | 13.5 (11.1)
  Change at Month 1 (n= 65) | 1.0 (8.6)
  Change at Month 2 (n= 62) | 1.5 (10.6)
  Change at Month 3 (n= 64) | -0.5 (9.9)
  Change at Month 4 (n= 58) | -1.0 (9.8)
  Change at Month 5 (n= 58) | -1.1 (8.6)
  Change at Month 6 (n= 56) | 0.9 (9.2)
  Change at Month 9 (n= 58) | 0.9 (10.7)
  Change at Month 12 (n= 57) | 1.6 (10.8)
  Change at Month 18 (n= 61) | -0.2 (9.0)
  Change at Month 24 (n= 63) | 0.1 (10.1)

7. Secondary Outcome: Change From Baseline in Center for State-trait Anger Expression Inventory 2 (STAXI-state) Score at Months 1, 2, 3, 4, 5, 6, 9, 12, 18 and 24
Description: STAXI-state scale measures the intensity of anger as an emotional state (state anger) and the disposition to experience angry feelings as a personality trait (trait anger). In this study only 1 of the original 6 scales was used, the state anger scale, which measures the intensity of anger at a given moment as emotional state. This scale consists of 15 items graded in 4 degrees from 1 (not at all) to 4 (very much), where 4 corresponds to the worst state. The total score range from 1 (not at all) to 60 (very much), where 60 corresponds to the worst state. (Spielberger CD, 1996)
Time Frame: Baseline, Months 1, 2, 3, 4, 5, 6, 9, 12, 18 and 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Interferon-beta
Number analyzed (Participants) | 70
units on a scale
  Baseline (n= 70) | 16.8 (4.1)
  Change at Month 1 (n= 65) | 0.0 (4.2)
  Change at Month 2 (n= 62) | 1.0 (5.3)
  Change at Month 3 (n= 64) | -0.0 (5.3)
  Change at Month 4 (n= 59) | -0.3 (4.7)
  Change at Month 5 (n= 58) | -0.0 (2.9)
  Change at Month 6 (n= 56) | 1.1 (7.6)
  Change at Month 9 (n= 58) | 1.1 (5.9)
  Change at Month 12 (n= 57) | 0.9 (5.7)
  Change at Month 18 (n= 61) | 0.8 (5.4)
  Change at Month 24 (n= 63) | 1.0 (5.5)

8. Secondary Outcome: Change From Baseline in Fatigue Score at Months 1, 2, 3, 6, 12 and 24
Description: Fatigue scale was derived from the United Kingdom Neurological Disability Scale (UKNDS), and evaluates fatigue according to the participant's subjective impression and the functional disability that it causes. 'Yes' or 'No' answers result in a score that ranges from 0 to 5, where a score 5 shows worse state. (Sharrack B et al., 1999)
Time Frame: Baseline, Months 1, 2, 3, 6, 12, and 24
Population: ITT population. 'N' (number of participants analyzed) signifies those participants who were evaluated for this measure. 'n' signifies those participants who were evaluated for this measure at that time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Interferon-beta
Number analyzed (Participants) | 62
units on a scale
  Baseline (n= 62) | 2.1 (1.7)
  Change at Month 1 (n= 58) | 0.5 (1.6)
  Change at Month 2 (n= 55) | 0.4 (1.5)
  Change at Month 3 (n= 56) | 0.2 (1.8)
  Change at Month 6 (n= 50) | 0.4 (1.8)
  Change at Month 12 (n= 49) | 0.1 (1.8)
  Change at Month 24 (n= 56) | -0.1 (2.1)

ADVERSE EVENTS:
Time Frame: Baseline to Month 24
Description: An adverse event (AE) was defined as any untoward medical occurrence in the form of signs, symptoms, abnormal laboratory findings, or diseases that emerges or worsens relative to baseline during a clinical study with an Investigational Medicinal Product (IMP), regardless of causal relationship and even if no IMP has been administered.
Arm/Group | Interferon-beta
Serious Adverse Events (participants affected / at risk) | 9/76
Other Adverse Events (participants affected / at risk) | 62/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Interferon-beta (N=76)
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sudden Hearing Loss (Ear and labyrinth disorders) | 1 (1)
Depression (Psychiatric disorders) | 3 (3)
Abortion (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Drug Dependence (Psychiatric disorders) | 1 (1)
Aggressivity (Psychiatric disorders) | 1 (1)
Suicide Attempt (Psychiatric disorders) | 1 (1)
Neck Injury (Injury, poisoning and procedural complications) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Interferon-beta (N=76)
Headache (Nervous system disorders) | 2 (2)
Multiple Sclerosis Relapse (Nervous system disorders) | 40 (40)
Migraine (Nervous system disorders) | 2 (2)
Carpal Tunnel Syndrome (Nervous system disorders) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1)
Nystagmus (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
Restless Legs Syndrome (Nervous system disorders) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1)
Influenza Like Illness (General disorders) | 18 (18)
Fatigue (General disorders) | 11 (11)
Injection Site Pain (General disorders) | 7 (7)
Injection Site Erythema (General disorders) | 5 (5)
Irritability (General disorders) | 2 (2)
Injection Site Haematoma (General disorders) | 1 (1)
Injection Site Reaction (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Depression (Psychiatric disorders) | 6 (6)
Anxiety (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2)
Depressed Mood (Psychiatric disorders) | 1 (1)
Emotional Distress (Psychiatric disorders) | 1 (1)
Mania (Psychiatric disorders) | 1 (1)
Panic Attack (Psychiatric disorders) | 1 (1)
Sleep Disorder (Psychiatric disorders) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2)
Influenza (Infections and infestations) | 2 (2)
Tonsillitis (Infections and infestations) | 2 (2)
Urinary Tract Infection (Infections and infestations) | 2 (2)
Acarodermatitis (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Rhinolaryngitis (Infections and infestations) | 1 (1)
Tracheitis (Infections and infestations) | 1 (1)
Urinary Tract Infection ba (Infections and infestations) | 1 (1)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Tendon Disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1)
Faecal Incontinence (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Ankle Fracture (Injury, poisoning and procedural complications) | 1 (1)
Clavicle Fracture (Injury, poisoning and procedural complications) | 1 (1)
Joint Dislocation (Injury, poisoning and procedural complications) | 1 (1)
Procedural Headache (Injury, poisoning and procedural complications) | 1 (1)
Upper Limb Fracture (Injury, poisoning and procedural complications) | 1 (1)
Wrist Fracture (Injury, poisoning and procedural complications) | 1 (1)
Deafness (Ear and labyrinth disorders) | 1 (1)
Menlere's Disease (Ear and labyrinth disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Cytolytic Hepatitis (Hepatobiliary disorders) | 3 (3)
Hepatitis (Hepatobiliary disorders) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Gamma-glutamyltransferase (Investigations) | 1 (1)
Liver Function Test Abnormal (Investigations) | 1 (1)
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)
Raynaud's Phenomenon (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other